CLINICAL TRIAL: NCT04790669
Title: Comparative Effects of Daily Adjustable Progressive Resistance Exercises Technique and Close Kinetic Chain Exercises on Extensor Lag in Post-operative Knee Stiffness
Brief Title: DAPRE Exercises Technique and CKC Exercises on Extensor Lag in Post Knee Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/021 Shanza Tanveer
Record Dates: First submitted 2021-03-06; First posted 2021-03-10 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Extensor Lag; Post-operative Knee Stiffness
Keywords: DAPRE; CKC exercises; Extensor lag
MeSH Terms: interventions — Conization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily adjustable progressive resistance exercises (DAPRE) (Experimental): DAPRE technique, hot pack, stretching exercises.
  Interventions: Procedure: Daily adjustable progressive resistance exercises (DAPRE)
- Close kinetic chain exercises (CKC). (Experimental): CKC exercises, hot pack, stretching exercises
  Interventions: Procedure: Close kinetic chain exercises (CKC).

INTERVENTIONS:
Procedure: Daily adjustable progressive resistance exercises (DAPRE) — Daily adjustable progressive resistance exercises (DAPRE) In Group A, 11 participants were received Conventional physiotherapy treatment in addition to DAPRE technique by leg extension machine. In DAPRE technique, four sets of exercises were performed. The first two sets of exercise consisted of ten and then six repetitions, per- formed against one-half and three-fourths of the previously established working weight. Working weight is the amount of weight a patient uses during an individual session. The full working weight was used on the third set, and the patient performed as many repetitions as possible. After performing each of the third and fourth sets, patients rested for 1 min.6 weeks (3 sessions per week)• Hot pack: 10 min• Stretching of calf and hamstring muscle: 10 min. Assessment was done via WOMAC index, universal goniometer, numeric pain rating scale & sphygmomanometer.
  Arms: Daily adjustable progressive resistance exercises (DAPRE)
Procedure: Close kinetic chain exercises (CKC). — Close kinetic chain exercises (CKC). In Group B, 11 participants was received Conventional physiotherapy treatment in addition to close kinetic chain exercises. Close kinetic chain exercises for extensor lag was seated leg press, double or single one third knee bend, step up and down exercise, wall slide with weight. Treatment time was 30 minutes and three session per week was applied on alternate day for up to 6 weeks. Pre interventional readings will be taken at baseline & post interventional readings at 6th week. 6 weeks (3 sessions per week) • Hot pack: 10 min • Stretching of calf and hamstring muscle: 10 min. Assessment was done via WOMAC index, universal goniometer, numeric pain rating scale & sphygmomanometer.
  Arms: Close kinetic chain exercises (CKC).

SUMMARY:
This project was a Randomized clinical trial conducted on extensor lag in post-operative knee stiffness patient to compare the effects of The Daily Adjustable Progressive Resistive Exercise (DAPRE) technique versus Close kinetic chain (CKC) exercise training in people who had undergone knee stiffness, m so that we can have best treatment option for patients with extensor lag.

DETAILED DESCRIPTION:
Probability Convenient sampling was done. Patients following eligibility criteria from Physiotherapy department of PSRD, Lahore, were considered. Sample size was calculated with Epi-tool calculator. 22 Participants were randomly allocated in two groups equally via convenient sampling method. Baseline assessment was done initially. Group A, 11 participants will receive Conventional physiotherapy treatment in addition to DAPRE technique by leg extension machine. In DAPRE technique, four sets of exercises were performed. The first two sets of exercise consisted of ten and then six repetitions, per- formed against one-half and three-fourths of the previously established working weight. Working weight is the amount of weight a patient uses during an individual session. The full working weight was used on the third set, and the patient performed as many repetitions as possible. After performing each of the third and fourth sets, patients rested for 1 min. 6 weeks (3 sessions per week)• Hot pack: 10 min• Stretching of calf and hamstring muscle: 10 min. Group B, 11 participants will receive Conventional physiotherapy treatment in addition to close kinetic chain exercises. Close kinetic chain exercises for extensor lag is seated leg press, double or single one third knee bend, step up and down exercise, wall slide with weight. Treatment time will be 30 minutes and three session per week will be applied on alternate day for up to 6 weeks. Pre interventional readings will be taken at baseline & post interventional readings at 6th week. 6 weeks (3 sessions per week) • Hot pack: 10 min • Stretching of calf and hamstring muscle: 10 min. All participants were provided written informed consent prior to commencement of the procedures. They were free to quit the treatment at any stage of research. Data was analyzed by using SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative knee stiffness (patients with 1-3 month stiffness).
* Both male and female , age 30-60 years.
* Willing to participate in research.

Exclusion Criteria:

Pre-operative knee stiffness

* Severe cardiopulmonary disease
* Patients undergoing chemotherapy
* Any traumatic injury/ Acute inflammatory muscular pathology
* TKR & hip pathology and replacement
* Meniscal tear

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Change in knee functional Improvement by WOMAC index | 6 weeks (3 sessions per week).
  By using WOMAC index, knee functional improvement was checked at baseline & post interventional readings at 6th week.
Change in knee range of motion by universal goniometer. | 6 weeks (3 sessions per week).
  Change in ROM at baseline & post interventional readings at 6th week.
Change in pain by 'Numeric Pain Rating Scale' | 6 weeks (3 sessions per week).
  Change in pain was measured at baseline & post interventional readings at 6th week.
Change in strength by Sphygmomanometer | 6 weeks (3 sessions per week).
  Change in strength was measured at baseline & post interventional readings at 6th week.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ardali G. A daily adjustable progressive resistance exercise protocol and functional training to increase quadriceps muscle strength and functional performance in an elderly homebound patient following a total knee arthroplasty. Physiother Theory Pract. 2014 May;30(4):287-97. doi: 10.3109/09593985.2013.868064. Epub 2014 Jan 7. PMID 24397371
- [Background] Wawrzyniak JR, Tracy JE, Catizone PV, Storrow RR. Effect of closed chain exercise on quadriceps femoris peak torque and functional performance. J Athl Train. 1996 Oct;31(4):335-40. PMID 16558420
- [Background] Knight KL. Quadriceps Strengthening with the DAPRE Technique: Case studies with Neurological Implications. J Orthop Sports Phys Ther. 1990;12(2):66-71. doi: 10.2519/jospt.1990.12.2.66. PMID 18787253